CLINICAL TRIAL: NCT06247488
Title: Randomized, Double-blind, Active & Placebo-controlled, 6-way Crossover Study of Abuse Potential of Oral Gabapentin Enacarbil IR Capsules With and Without Oxycodone in Healthy, Nondependent, Recreational Opioid Users
Brief Title: Abuse Potential of HORIZANT With and Without Oxycodone in Healthy, Nondependent Recreational Opioid Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: AR26.3031.2
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Abuse Potential
MeSH Terms: interventions — Oxycodone; 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): oral masked Placebo
  Interventions: Drug: Placebo
- Oxycodone 20 mg (Active Comparator): oral active control
  Interventions: Drug: Oxycodone 20 mg
- GE-IR 200mg (Experimental): single oral dose
  Interventions: Drug: GE-IR 200 mg
- GE-IR 450 mg (Experimental): single oral dose
  Interventions: Drug: GE-IR 450 mg
- GE-IR 200 mg + Oxycodone 20 mg (Experimental): oral doses given together
  Interventions: Drug: Oxycodone 20 mg; Drug: GE-IR 200 mg
- GE-IR 450 mg + Oxycodone 20 mg (Experimental): oral doses given together
  Interventions: Drug: Oxycodone 20 mg; Drug: GE-IR 450 mg

INTERVENTIONS:
Drug: Placebo — Participant will receive oral dose of placebo.
  Other Names: matching over-encapsulated capsule
  Arms: Placebo
Drug: Oxycodone 20 mg — Participant will receive oral dose of oxycodone 20 mg.
  Other Names: Oxycontin
  Arms: GE-IR 200 mg + Oxycodone 20 mg; GE-IR 450 mg + Oxycodone 20 mg; Oxycodone 20 mg
Drug: GE-IR 200 mg — Participant will receive oral dose of GE-IR 200 mg and oxycodone 20 mg.
  Other Names: Gabapentin Enacarbil, Horizant
  Arms: GE-IR 200 mg + Oxycodone 20 mg; GE-IR 200mg
Drug: GE-IR 450 mg — Participant will receive oral dose of GE-IR 450 mg and oxycodone 20 mg.
  Other Names: Gabapentin Enacarbil, Horizant
  Arms: GE-IR 450 mg; GE-IR 450 mg + Oxycodone 20 mg

SUMMARY:
The purpose of this study is to assess the abuse potential of gabapentin enacarbil immediate release capsules taken alone and in combination with oxycodone in healthy adult, non-dependent, recreational opioid users.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the abuse potential of gabapentin enacarbil immediate-release (GE-IR), the active moiety in Horizant, taken alone and taken in combination with oxycodone, compared to that of oxycodone alone.

This study is a randomized, double-blind, active- and placebo-controlled, 6-way crossover design, aimed to assess the abuse potential, safety, and pharmacokinetics (PK) of GE-IR doses when administered alone or in combination with an opioid active control (oxycodone), and compared to placebo and oxycodone intake alone, in healthy, nondependent, recreational opioid users.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF),
2. Stated willingness to comply with all study procedures and availability for the duration of the study,
3. Male or female, between 18 and 55 years of age, inclusive,
4. Current nondependent, recreational opioid user who has used opioid drugs for recreational (nontherapeutic) purposes (i.e., for psychoactive effects) at least 5 times in the subject's lifetime and at least once in the last 12 weeks,
5. Body mass index (BMI) within 18.0 kg/m2 to 36.0 kg/m2, inclusive,
6. If female, meets 1 of the following criteria:

   1. If of childbearing potential agrees to use 1 of the accepted contraceptive regimens from at least 30 days prior to the first study treatment administration, during the study, and for at least 30 days after the last dose of the study treatment. An acceptable method of contraception includes 1 of the following:

      * Abstinence from heterosexual intercourse,
      * Hormonal contraceptives (birth control pills, injectable/implantable/insertable hormonal birth control products, transdermal patch), or
      * Intrauterine device (IUD; with or without hormones). Or
   2. If of childbearing potential agrees to use a double barrier method (e.g., condom and spermicide) during the study and for at least 30 days after the last dose of study treatment.

      Or
   3. If of non-childbearing potential, defined as surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy or tubal ligation) or is in a postmenopausal state (i.e., at least 1 year without menses without an alternative medical condition and confirmed follicle stimulating hormone (FSH) ≥ 40 milli-International unit (mIU)/mL prior to the first study treatment administration),
7. If male and engaging in sexual activity that has the risk of pregnancy must agree to use a double barrier method (e.g., condom and spermicide) and agree to not donate sperm during the study and for at least 90 days after the last dose of study treatment, a male who has a pregnant partner shall be excluded,
8. Healthy, as determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs or clinical laboratory (including hematology, clinical chemistry, urinalysis, and serology [screening visit only]) at screening visit and admission, in the opinion of an investigator.
9. Negative COVID-19 test prior to each admission.

Exclusion Criteria:

1. History of significant hepatic, renal, cardiovascular, pulmonary, hematologic, neurological, psychiatric, gastrointestinal, endocrine, immunologic, ophthalmologic, or dermatologic disease of any etiology (including infections),
2. Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability with the exception that cholecystectomy is permitted at the discretion of an investigator,
3. Presence of any significant respiratory illness or presence or history of chronic respiratory disease (e.g., upper respiratory illness, sleep apnea, emphysema, asthma) at screening (subjects with acute respiratory illness may be rescheduled upon resolution at the discretion of an investigator),
4. Personal or family history (first degree relatives) of allergy, hypersensitivity, or drug rash with eosinophilia and systemic symptoms (DRESS) syndrome to gabapentin enacarbil,gabapentin or any drug product including naloxone, opioids (e.g., oxycodone), or related drugs or known excipients of any of the drug products in this study (e.g. lactose),
5. History of sensitivity to or poor tolerance of gabapentin enacarbil, gabapentin, pregabalin, naloxone, or oxycodone,
6. Female who is lactating at screening,
7. Female who is pregnant according to the pregnancy test at screening or prior to the first study treatment administration or planning to become pregnant within 30 days following the last study treatment administration,
8. History of substance or alcohol dependence (excluding nicotine and caffeine) within the past 2 years, as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV), and/or subject has ever been in a drug or alcohol rehabilitation program within the last 2 years,
9. Subjects with positive urine drug screen (UDS) results at screening and admission will be assessed for inclusion at the discretion of an Investigator. If tetrahydrocannabinol (THC) is positive at admission to the qualification phase and treatment phase, a cannabis intoxication evaluation will be done by an investigator and subjects may be permitted to continue in the study, rescheduled, or discontinued at the discretion of an investigator. Other positive test results should be reviewed to determine if the subject may be rescheduled, in the opinion of the investigator,
10. Is a heavy smoker (>20 cigarettes per day or nicotine-equivalent) and/or is unable to abstain from smoking or unable to abstain from the use of prohibited nicotine-containing products for at least 1 hour before and 6 hours after study treatment administration (including e-cigarettes, pipes, cigars, chewing tobacco, nicotine topical patches, nicotine gum, or nicotine lozenges),
11. Is a heavy opioid user and not likely to be sensitive to a 20 mg dose of oxycodone, in the opinion of an investigator or designee,
12. Regularly consumes excessive amounts of caffeine or xanthines within 30 days prior to screening, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day,
13. History of suicidal ideation or suicidal behaviour within 2 years of screening, showing suicidal tendency as per the Columbia Suicide Severity Rating Scale (C-SSRS) administered at screening, or is currently at risk of suicide in the opinion of an investigator,
14. Presence of clinically significant ECG abnormalities at the screening visit, as defined by medical judgment, Note: QT corrected according to Fridericia's formula (QTcF) interval of >450 msec in male subjects or >470 msec in female subjects will be exclusionary. The ECG may be repeated once for confirmatory purposes if the initial value obtained exceeds the limits specified,
15. Has creatinine clearance ≤60ml/min as calculated by the Cockcroft-Gault equation,
16. Any history of tuberculosis,
17. Positive screening results to human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B virus surface antigen (HBsAg) or hepatitis C virus antibody (HCVAb) tests,
18. Intake of an investigational product (IP) within 30 days or 5 times the half-life (whichever is longer) prior to screening,
19. Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) in the 30 days prior to the first study treatment administration, that in the opinion of an investigator would put into question the status of the subject as healthy,
20. Use of over-the-counter (OTC) products (including herbal preparations and supplements) within 7 days prior to the first study treatment administration, with the exception of ibuprofen or acetaminophen,
21. Use of a prohibited medication as specified in section 4.7,
22. Donation of plasma in the 7 days prior to screening,
23. Blood donation (excluding plasma) of approximately 500 mL of blood in the 56 days prior to screening,
24. Is, in the opinion of an investigator or designee, considered unsuitable or unlikely to comply with the study protocol for any reason.
25. Poor venous access at screening, as judged by an investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Clinical Kansas, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 110 volunteers consented for the study and entered into a qualification phase.
Pre-assignment Details: In the qualification phase subjects were given a naloxone challenge to rule out drug dependent participants. Those that passed the challenge were randomized to get crossover doses of placebo and Oxycodone in random order to ensure they could tolerate and detect the effects of Oxy. 72 subjects completed qualification and 9 of those did not proceed to the treatment phase. 63 started the treatment phase and got at least one dose of study drug. 54 completed and were analyzed.
Groups:
- ABFCED: Period 1 Placebo, Period 2 Oxycodone (Oxy) 20mg, Period 3 Gabapentin Enacarbil Immediate Release (GE-IR) 450mg, Period 4 GE-IR 200mg + Oxy 20mg, Period 5 GE-IR 200mg, Period 6 GE-IR 450 + Oxy 20mg
- BCADFE: Period 1 Oxy 20 mg, Period 2 GE-IR 200mg + Oxy 20mg, Period 3 Placebo, Period 4 GE-IR 450 + Oxy 20mg, Period 5 GE-IR 450 mg, Period 6 GE-IR 200
- CBDEAF: Period 1 GE-IR 200mg + Oxy 20mg, Period 2 GE-IR 450 + Oxy 20mg, Period 3 Oxy 20 mg, Period 4 GE-IR 200mg. Period 5 Placebo, Period 6 GE-IR 450
- DECFBA: Period 1 GE-IR 450 + Oxy 20mg, Period 2 GE-IR 200 mg, Period 3 GE-IR 200 mg + Oxy 20mg, Period 4 GE-IR 450 mg, Period 5 Oxy 20 mg, Period 6 Placebo
- EFDACB: Period 1 GE-IR 200 mg, Period 2 GE-IR 450 mg, Period 3 GE-IR 450 mg + 20 mg Oxy, Period 4 Placebo, Period 5 GE-IR 200 mg + Oxy 20 mg, Period 6 Oxy 20 mg
- FAEBDC: Period 1 GE-IR 450 mg, Period 2 Placebo, Period 3 GE-IR 200 mg, Period 4 Oxy 20 mg, Period 5 GE-IR 450 mg + 20 mg Oxy, Period 6 GE-IR 200 mg + Oxy 20 mg
Period: First Intervention (1 Day)
Arm/Group | ABFCED | BCADFE | CBDEAF | DECFBA | EFDACB | FAEBDC
Started | 10 | 10 | 11 | 12 | 10 | 10
Completed | 10 | 10 | 11 | 12 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First Washout (3 Days)
Arm/Group | ABFCED | BCADFE | CBDEAF | DECFBA | EFDACB | FAEBDC
Started | 10 | 10 | 11 | 12 | 10 | 10
Completed | 10 | 10 | 11 | 12 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | ABFCED | BCADFE | CBDEAF | DECFBA | EFDACB | FAEBDC
Started | 10 | 10 | 11 | 12 | 10 | 10
Completed | 10 | 10 | 11 | 12 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout From 2nd Dose (3 Days)
Arm/Group | ABFCED | BCADFE | CBDEAF | DECFBA | EFDACB | FAEBDC
Started | 10 | 10 | 11 | 12 | 10 | 10
Completed | 9 | 10 | 11 | 11 | 10 | 10
Not Completed | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | ABFCED | BCADFE | CBDEAF | DECFBA | EFDACB | FAEBDC
Started | 9 | 10 | 11 | 11 | 10 | 10
Completed | 9 | 10 | 11 | 11 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout of Third Dose (3 Days)
Arm/Group | ABFCED | BCADFE | CBDEAF | DECFBA | EFDACB | FAEBDC
Started | 9 | 10 | 11 | 11 | 10 | 10
Completed | 8 | 10 | 11 | 11 | 10 | 10
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention (One Day)
Arm/Group | ABFCED | BCADFE | CBDEAF | DECFBA | EFDACB | FAEBDC
Started | 8 | 10 | 11 | 11 | 10 | 10
Completed | 8 | 10 | 11 | 11 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout of Fourth Dose (3 Days)
Arm/Group | ABFCED | BCADFE | CBDEAF | DECFBA | EFDACB | FAEBDC
Started | 8 | 10 | 11 | 11 | 10 | 10
Completed | 8 | 10 | 11 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Period: Fifth Intervention (1 Day)
Arm/Group | ABFCED | BCADFE | CBDEAF | DECFBA | EFDACB | FAEBDC
Started | 8 | 10 | 11 | 10 | 10 | 10
Completed | 8 | 10 | 11 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout of 5th Dose (3 Days)
Arm/Group | ABFCED | BCADFE | CBDEAF | DECFBA | EFDACB | FAEBDC
Started | 8 | 10 | 11 | 10 | 10 | 10
Completed | 8 | 9 | 10 | 10 | 10 | 7
Not Completed | 0 | 1 | 1 | 0 | 0 | 3
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Period: Sixth Intervention (1 Day)
Arm/Group | ABFCED | BCADFE | CBDEAF | DECFBA | EFDACB | FAEBDC
Started | 8 | 9 | 10 | 10 | 10 | 7
Completed | 8 | 9 | 10 | 10 | 10 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subject who passed the naloxone challenge (showing no signs of withdrawal and could distinguish oxycodone from placebo in a blinded qualification test where subjects got both treatments over two days in a random order.
Groups:
- Subjects Eligible for Treatment Phase: Subjects that met all eligibility and qualification criteria and entered the study treatment phase.
Arm/Group | Subjects Eligible for Treatment Phase
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 51
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 63
Opioid Use in the Past 12 Months [Mean (Full Range); unit: uses] | 12 [1 to 69]

OUTCOME MEASURES:

1. Primary Outcome: Drug Liking Visual Analog Scale (VAS)
Description: Mean difference in Drug Liking Emax over 24 hours for Drug Liking ("At this moment, my liking for this drug is"), assessed on a bipolar (0 to 100 points; 0: Strong disliking, 50: Neither like nor dislike, 100: Strong liking) VAS.
Time Frame: approximately 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, and 24 hours postdose in the treatment phase and per period of the treatment phase
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- GE-IR 200 mg + Oxycodone 20 mg: oral doses given together
  : Participant will receive oral dose of oxycodone 20 mg.
  GE-IR 200 mg: Participant will receive oral dose of GE-IR 200 mg and oxycodone 20 mg.
- GE-IR 450 mg + Oxycodone 20 mg: oral doses given together
  Participant will receive oral dose of oxycodone 20 mg.
  GE-IR 450 mg: Participant will receive oral dose of GE-IR 450 mg and oxycodone 20 mg.
Arm/Group | Placebo | Oxycodone 20 mg | GE-IR 200mg | GE-IR 450 mg | GE-IR 200 mg + Oxycodone 20 mg | GE-IR 450 mg + Oxycodone 20 mg
Number analyzed (Participants) | 54 | 54 | 54 | 54 | 54 | 54
score on a scale | 56.4 (1.75) | 84.9 (2.08) | 59.6 (2.28) | 64.6 (2.45) | 84.5 (2.11) | 86.6 (2.03)

2. Secondary Outcome: Overall Drug Liking VAS
Description: Mean difference in Emax for Overall Drug Liking ("Overall, my liking for this drug is"), assessed on a bipolar (0 to 100 points; 0: Strong disliking, 50: Neither like nor dislike, 100: Strong liking) VAS.
Time Frame: Approximately 12 and 24 hours postdose in the treatment phase and per period of the treatment phase
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Oxycodone 20 mg | GE-IR 200mg | GE-IR 450 mg | GE-IR 200 mg + Oxycodone 20 mg | GE-IR 450 mg + Oxycodone 20 mg
Number analyzed (Participants) | 54 | 54 | 54 | 54 | 54 | 54
score on a scale | 60.3 (2.33) | 85.6 (2.08) | 57.5 (2.03) | 65.2 (2.66) | 82.4 (2.51) | 84.5 (2.66)

3. Secondary Outcome: Take Drug Again VAS
Description: Mean difference in Emax for Take Drug Again ("I would take this drug again"), assessed on a bipolar (0 to 100 points; 0: Definitely would not 50: Neither would nor would not, 100: Definitely would) VAS.
Time Frame: Approximately 12 and 24 hours postdose in the treatment phase and per period of the treatment phase
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Oxycodone 20 mg | GE-IR 200mg | GE-IR 450 mg | GE-IR 200 mg + Oxycodone 20 mg | GE-IR 450 mg + Oxycodone 20 mg
Number analyzed (Participants) | 54 | 54 | 54 | 54 | 54 | 54
score on a scale | 60.8 (2.47) | 85.9 (2.25) | 56.7 (2.23) | 65.9 (2.69) | 85.2 (2.41) | 85.9 (2.67)

4. Secondary Outcome: High VAS
Description: Mean difference in Emax for High ("At this moment, I'm feeling high"), assessed on a unipolar (0 to 100 points; 0: Not at all, 100: Extremely) VAS.
Time Frame: within 1 hour prior to and approximately 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, and 24 hours postdose in the treatment phase and per period of the treatment phase
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Oxycodone 20 mg | GE-IR 200mg | GE-IR 450 mg | GE-IR 200 mg + Oxycodone 20 mg | GE-IR 450 mg + Oxycodone 20 mg
Number analyzed (Participants) | 54 | 54 | 54 | 54 | 54 | 54
score on a scale | 8.6 (2.72) | 66.3 (4.20) | 10.5 (3.24) | 20.1 (4.00) | 65.1 (4.02) | 73.2 (3.46)

ADVERSE EVENTS:
Time Frame: AEs were monitored through the 3-day qualification phase, and throughout the 17-day treatment phase until the final follow-up visit at day 23 (+/- 2 days).
Arm/Group | Placebo | Oxycodone 20 mg | GE-IR 200mg | GE-IR 450 mg | GE-IR 200 mg + Oxycodone 20 mg | GE-IR 450 mg + Oxycodone 20 mg
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61 | 0/60 | 0/60 | 0/57 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61 | 0/60 | 0/60 | 0/57 | 0/61
Other Adverse Events (participants affected / at risk) | 12/61 | 24/61 | 8/60 | 16/60 | 28/57 | 33/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=61) | Oxycodone 20 mg (N=61) | GE-IR 200mg (N=60) | GE-IR 450 mg (N=60) | GE-IR 200 mg + Oxycodone 20 mg (N=57) | GE-IR 450 mg + Oxycodone 20 mg (N=61)
Euphoric Mood (Psychiatric disorders) | 2 (2) | 10 (10) | 2 (2) | 7 (7) | 11 (11) | 19 (19)
Somnolence (Nervous system disorders) | 6 (6) | 4 (4) | 1 (1) | 3 (3) | 8 (8) | 11 (11)
headache (Nervous system disorders) | 1 (1) | 2 (3) | 1 (1) | 5 (5) | 3 (3) | 1 (1)
puritis (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 7 (7) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Emotional Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dizzyness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling of Relaxation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Feeling Hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Noncardiac Chestpain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
backpain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
anaphylactoid reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
63 subjects entered the treatment phase and were assessed for adverse events. 11 discontinued over the course of the 6 study periods. 54 subjects were part of the analysis population. This met the study goal for population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT06247488/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT06247488/SAP_001.pdf